CLINICAL TRIAL: NCT03086070
Title: Omeprazole 20 mg in Patients With Laryngopharyngeal reﬂux and Comorbid Chronic Rhinosinusitis - a Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Omeprazole 20 mg in Patients With Laryngopharyngeal reﬂux and Comorbid Chronic Rhinosinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Srebrnjak (Other)
Collaborators: University Hospital Center Sisters of Charity, Zagreb, Croatia (Unknown); Belupo (Other)
Responsible Party: Principal Investigator, Davor Plavec, Assoc.Prof., MD, PhD, Children's Hospital Srebrnjak
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS-ENT01
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Laryngopharyngeal Reflux; Chronic Rhinosinusitis (Diagnosis)
Keywords: omeprazole; placebo; treatment; adults
MeSH Terms: conditions — Laryngopharyngeal Reflux; Disease | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): omeprazole 20 mg capsule once daily for 8 weeks
  Interventions: Drug: Omeprazole 20mg
- Placebo arm (Placebo Comparator): matching placebo capsules ones daily for 8 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Omeprazole 20mg — omeprazole 20 mg capsules were administered per os half an hour before breakfast for 8 weeks
  Arms: Treatment arm
Drug: Placebo oral capsule — Matching placebo oral capsules were administered per os half an hour before breakfast for 8 weeks
  Arms: Placebo arm

SUMMARY:
The hypothesis of this study is that a gastroesophageal reflux recommended treatment with proton pump inhibitor (dose and duration) compared to placebo significantly reduces both the signs and symptoms of laryngopharyngeal reﬂux and comorbid chronic rhinosinusitis. Primary objective was to determine whether 8 weeks of treatment with omeprazole 20 mg ones daily (OD) significantly reduces the signs and symptoms of laryngopharyngeal reﬂux when compared to placebo in patients with laryngopharyngeal reﬂux with comorbid chronic rhinosinusitis. Secondary objectives were to determine whether 8 weeks of treatment with omeprazole 20 mg OD significantly reduces the signs and symptoms of comorbid chronic rhinosinusitis in patients with laryngopharyngeal reﬂux when compared to matching placebo; and to investigate the association of the severity of signs and symptoms of laryngopharyngeal reﬂux with the ones of chronic rhinosinusitis in the same group of patients. The research was carried out as a double blind randomized placebo controlled trial. Patients were randomized into two groups in an approximate 1:1 ratio using a concealed random sequence. After randomization and initial assessment treatment was initialized. Patients on active treatment were given omeprazole 20 mg once daily half an hour before breakfast for 8 weeks, while those in the placebo group were given matching placebo tablets using the same regimen for 8 weeks as the group on the active treatment. Patients were reassessed at the end of treatment for signs and symptoms of laryngopharyngeal reﬂux and comorbid chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* laryngopharyngeal reﬂux
* chronic rhinosinusitis

Exclusion Criteria:

* allergic rhinitis
* asthma
* cystic fibrosis
* nasal polyposis
* severe systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in signs and symptoms of laryngopharyngeal reﬂux | 8 weeks
  Reﬂux symptom index (RSI) score
Reduction in signs and symptoms of laryngopharyngeal reﬂux | 8 weeks
  Reﬂux finding score (RFS)

SECONDARY OUTCOMES:
Reduction of signs and symptoms of comorbid chronic rhinosinusitis | 8 weeks
  Nasal obstruction, anterior/posterior nasal drip, headache, sneezing, cough, smell and taste disorder with frequency and intensity of the symptoms was graded from 0 (no problem) to 3 (severe problem).
  Nasal endoscopy with endoscopy scores were based on the assessment of nasal mucosa edema, secretions and presence of polyps and were graded from 0 (no problem) to 3 (severe problem).
Association of the severity of signs and symptoms of laryngopharyngeal reﬂux with the ones of chronic rhinosinusitis | Baseline and after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Srđan A Anzić, MD, PhD, Principal Investigator — Children's Hospital Srebrnjak

IPD SHARING:
Plan to Share IPD: No
Anonymised individual participant data can be obtained for other researchers on a written request to the principal investigator.

REFERENCES:
- [Result] Anzic SA, Turkalj M, Zupan A, Labor M, Plavec D, Baudoin T. Eight weeks of omeprazole 20 mg significantly reduces both laryngopharyngeal reflux and comorbid chronic rhinosinusitis signs and symptoms: Randomised, double-blind, placebo-controlled trial. Clin Otolaryngol. 2018 Apr;43(2):496-501. doi: 10.1111/coa.13005. Epub 2017 Oct 23. PMID 29024410